CLINICAL TRIAL: NCT06614010
Title: Effect of Different Administration Routes of Dexmedetomidine Combined with Ultrasound-Guided Fascia Iliaca Block on Emergence Agitation After Hip Replacement Surgery
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Pengcai Shi, Chief physician，Master Tutor, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LI
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Dexmedetomidine; Fascia Iliaca Block
Keywords: Fascia Iliaca Block; Dexmedetomidine; Emergence Agitation; Ropivacaine; Analgesic Mechanism
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group S1 (Experimental): Before anesthesia induction, an iliac fascia block was administered using 0.375% ropivacaine (30 mL) under ultrasound guidance, followed by conventional anesthesia induction. During the anesthesia maintenance phase, dexmedetomidine was infused intravenously at a rate of 0.5 µg/kg/h.
  Interventions: Drug: Dexmedetomidine Injection
- Group S2 (Experimental): Before anesthesia induction, an iliac fascia block was administered using a mixture of 0.375% ropivacaine and 1ug/kg dexmedetomidine (30ml) under ultrasound guidance. During the anesthesia maintenance phase, an equivalent volume of 0.9% sodium chloride injection was infused intravenously.
  Interventions: Drug: Ropivacaine and Dexmedetomidine
- Group C (Active Comparator): Before anesthesia induction, an iliac fascia block was performed using 0.375% ropivacaine (30 mL) under ultrasound guidance, followed by conventional anesthesia induction. During the anesthesia maintenance phase, an equivalent volume of 0.9% sodium chloride injection was infused intravenously.
  Interventions: Drug: Sodium Chloride Injection

INTERVENTIONS:
Drug: Dexmedetomidine Injection — Before anesthesia induction, an iliac fascia block was administered using 0.375% ropivacaine (30 mL) under ultrasound guidance, followed by conventional anesthesia induction. During the anesthesia maintenance phase, dexmedetomidine was infused intravenously at a rate of 0.5 µg/kg/h.
  Arms: Group S1
Drug: Ropivacaine and Dexmedetomidine — Before anesthesia induction, an iliac fascia block was administered using a mixture of 0.375% ropivacaine and 1ug/kg dexmedetomidine (30ml) under ultrasound guidance. During the anesthesia maintenance phase, an equivalent volume of 0.9% sodium chloride injection was infused intravenously.
  Arms: Group S2
Drug: Sodium Chloride Injection — Before anesthesia induction, an iliac fascia block was performed using 0.375% ropivacaine (30 mL) under ultrasound guidance, followed by conventional anesthesia induction. During the anesthesia maintenance phase, an equivalent volume of 0.9% sodium chloride injection was infused intravenously.
  Arms: Group C

SUMMARY:
To examine the impact of various administration routes of dexmedetomidine in conjunction with ultrasound-guided fascia iliaca block (FIB) on emergence agitation (EA) during the postoperative recovery period after hip replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 65 years, with no restriction on gender
2. diagnosis of hip joint disease necessitating hip arthroplasty
3. ASA grade I-II
4. no significant cardiopulmonary, hepatic, or renal dysfunction prior to the operation
5. no history of psychiatric disorders or long-term use of sedative medications prior to the operation
6. signing of an informed consent form to voluntarily participate in the study.

Exclusion Criteria:

1. patients allergic to or with contraindications to ropivacaine or dexmedetomidine
2. patients exhibiting symptoms of agitation or delirium prior to the procedure
3. patients with severe central or peripheral nervous system disorders
4. patients with coagulation disorders or receiving anticoagulant therapy
5. pregnant or breastfeeding women
6. patients who received other medications or treatments prior to the procedure that might affect the study results
7. patients unable to cooperate with the study or intolerant to ultrasound-guided iliofascial block

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Estimated)
Dates: Start 2023-02-05 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of awakening agitation | postoperative awakening period (1 min, 10 min, 20 min) and at the time of discharge from the PACU
  Riker sedation-agitation scale (SAS) scores were recorded at various time points during the postoperative awakening period (1 min, 10 min, 20 min) and at the time of discharge from the PACU for each group. These scores were used to evaluate the sedation and agitation status of the patients.

SECONDARY OUTCOMES:
Analgesic effect | postoperative awakening period (1 min, 10 min, 20 min) and at the time of discharge from the PACU
  The analgesic effect was recorded at various time points during the postoperative awakening period (1 min, 10 min, 20 min) and at the time of discharge from the PACU for each group. Analgesia was assessed using the Numerical Rating Scale (NRS), which ranges from 0 to 10, with higher scores indicating more severe pain.
Ramesay score | postoperative awakening period (1 min, 10 min, 20 min) and at the time of discharge from the PACU
  The sedation effect of patients in each group was recorded at various time points during the postoperative awakening period (1 min, 10 min, 20 min) and at the time of discharge from the PACU. Sedation was assessed using the Ramsay scale, which consists of 6 grades, with higher scores indicating deeper levels of sedation.
Hemodynamic parameters | During operation
  Comparisons of hemodynamic parameters among the three groups were made at several time points: after admission (T0), upon completion of anesthesia induction (T1), at the start of surgery (T2), one hour into the surgery (T3), at the end of surgery (T4), and at the removal of the laryngeal mask (T5). The parameters assessed included changes in systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate (HR), and oxygen saturation (SpO2).
Record of laryngeal mask removal time and adverse reactions | Within 24 hours after surgery
  The time of laryngeal mask removal was documented in detail for all three patient groups. Additionally, attention was given to monitoring and recording any adverse reactions occurring during the perioperative period.

CONTACTS AND LOCATIONS:
Locations (1):
- Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No